CLINICAL TRIAL: NCT07321457
Title: Effects of Watson's Human Caring Theory-Based Nursing Care on Fear of Childbirth and Birth Experience: A Randomized Controlled Trial
Brief Title: Effects of Watson's Human Caring Theory-Based Nursing Care on Fear of Childbirth and Birth Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Candan Ozturk, Co-Investigator, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YTK.1.01
Record Dates: First submitted 2025-12-15; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Fear of Childbirth; Childbirth Experience
Keywords: childbirth; caring; fear; nursing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Mothers in the intervention group received nursing care based on Watson's Human Caring Theory during labor. This care included emotional support, therapeutic communication, and individualized interventions aimed at reducing fear of childbirth and improving overall birth experience.
  Interventions: Behavioral: Intervention Group: Watson's Human Caring Theory-Based Nursing Care
- Control Group (Active Comparator): Mothers in the control group received routine nursing care during labor. No additional interventions based on Watson's Human Caring Theory were administered.
  Interventions: Behavioral: Routine Nursing Care

INTERVENTIONS:
Behavioral: Intervention Group: Watson's Human Caring Theory-Based Nursing Care — Mothers in the intervention group received nursing care based on Watson's Human Caring Theory during labor. This care included individualized emotional support, therapeutic communication, and other nursing interventions designed to reduce fear of childbirth and enhance overall birth experience. The program was specifically tailored to each mother's needs, distinguishing it from routine nursing care provided in standard labor management.
  Arms: Intervention Group
Behavioral: Routine Nursing Care — Mothers in the control group received routine nursing care during labor. No additional interventions based on Watson's Human Caring Theory were administered. This care followed standard hospital procedures for labor and delivery, without any individualized behavioral or supportive programs.
  Arms: Control Group

SUMMARY:
The purpose of this clinical trial was to evaluate the effect of integrating a nursing care program based on Watson's Theory of Human Caring into the childbirth process on mothers' fear of childbirth and childbirth experience among women who had uncomplicated vaginal births.

The study aimed to examine whether nursing care structured according to Watson's Theory of Human Caring differed from routine nursing care in terms of fear of childbirth and childbirth experience during labor.

Researchers compared an intervention group, which received Watson's Theory-based nursing care, with a control group, which received routine nursing care, using standardized assessment tools.

Participants:

Received either nursing care based on Watson's Theory of Human Caring or routine nursing care during labor

Completed the Fear of Childbirth Scale (FOBS) and the Questionnaire for Assessing Childbirth Experience (QACE)

Were monitored and assessed throughout the labor process

DETAILED DESCRIPTION:
This randomized controlled trial was designed to evaluate the effect of integrating a nursing care program based on Watson's Theory of Human Caring into the childbirth process on mothers' fear of childbirth and childbirth experience.

The study was conducted at a public hospital in Northern Cyprus between May 2024 and March 2025. A total of 30 mothers who experienced uncomplicated vaginal births were enrolled and randomly assigned to either the intervention group (n = 15) or the control group (n = 15).

The control group received routine nursing care, while the intervention group received nursing care structured according to Watson's Theory of Human Caring. The study employed a single-blind design, in which participants were unaware of their group allocation.

Data were collected using the Fear of Childbirth Scale (FOBS) and the Questionnaire for Assessing the Childbirth Experience - Short Version (QACE). These instruments were used to assess fear of childbirth and childbirth experience during labor and the postpartum period.

Statistical analyses were planned to compare outcomes between the intervention and control groups and to examine the effect of theory-based nursing care on fear of childbirth and childbirth experience.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ≥18 years, at 37-41 weeks of gestation, Pregnant women in the active phase of labor (cervical dilation ≥ 3 cm). Pregnant women who presented with spontaneous labor were directed to vaginal de-livery after physician evaluation.

Pregnant women carrying a single fetus in a vertex presentation. Pregnant women with an estimated fetal weight between 2500 4000 grams. Pregnant women undergo regular uterine contractions characteristic of the active phase.

Pregnant women who are literate in Turkish.

Exclusion Criteria:

* Pregnant women younger than 18 years. Pregnant women older than 45 years. Pregnant women with multiple pregnancies. Pregnant women with a history of in vitro fertilization (IVF). Pregnant women in the latent phase with cervical dilation < 3 cm. Pregnant women who received spinal, epidural, or general anesthesia during la-bor.

Pregnant women with a previous cesarean section (C/S). Pregnant women with a history of uterine surgery. Pregnant women whose delivery resulted in an emergency cesarean section. Pregnant women diagnosed with a mental disorder. Pregnant women showing signs of tokophobia (clinical fear of childbirth. Pregnant women who were separated from their newborn baby for medical reasons after delivery.

Pregnant women with a history of preeclampsia. Pregnant women with premature rupture of membranes (PROM). Pregnant women with placenta anomalies (placenta previa, placental abruptio, etc.).

Pregnant women with chronic diseases (DM, HT, etc.). Pregnant women with infectious diseases or active infections. Pregnant women with anemia. Pregnant women with fetal macrosomia. Pregnant women with vaginal bleeding. Pregnant women with abnormal vital signs. Pregnant women with presentation anomalies (breech, transverse)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who are biologically female and capable of giving birth were eligible to participate. There were no restrictions based on self-identified gender.
Enrollment: 30 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Birth Experience | 1-1.5 months postpartum
  Mothers' overall childbirth experience was assessed using the validated Questionnaire for Assessing Childbirth Experience - Short Version (QACE) through telephone interviews conducted 1 to 1.5 months after delivery. Each dimension of the QACE is scored on a scale ranging from 1 to 4, with higher scores indicating more negative childbirth experiences.
Fear of Childbirth Scale | During the active and transition phases of the first stage of labor
  The level of fear experienced by mothers during labor was assessed using the validated Fear of Childbirth Scale (FOBS). The total score of the FOBS ranges from 0 to 100, with higher scores indicating higher levels of fear of childbirth. A cut-off score of 50 was used to classify participants as having fear of childbirth.

CONTACTS AND LOCATIONS:
Overall Officials: Candan Ozturk, Prof. Dr., Principal Investigator — Near East University
Locations (1):
- Burhan Nalbantoglu state hospital, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared. The dataset contains sensitive personal health information collected from mothers during labor, and sharing is restricted to protect participant privacy and confidentiality.